CLINICAL TRIAL: NCT02699242
Title: Does Training on a Virtual Reality Bronchoscopy Simulator Improve Performance of Bronchoscopic Intubation in Patients?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, David Wong, Anesthesiologist, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 13-6321-BE
Record Dates: First submitted 2016-02-14; First posted 2016-03-04 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Endotracheal Intubation
Keywords: Fiberoptic intubation Training Simulation Performance

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simulator arm (Experimental): In the Simulation arm group the subjects will be trained on the virtual reality bronchoscopic simulator (ORSIM simulator) for up to 60 minutes as active intervention, before they undertake the 2nd Fiber optic intubations.
  Interventions: Device: Simulator (ORSIM) training
- Control arms (No Intervention): The control arm will be exposed only to the didactic teaching. The subjects will not undergo simulator training before undergoing 2nd fiber optic intubations.

INTERVENTIONS:
Device: Simulator (ORSIM) training — The simulator/intervention group will undergo training on the virtual reality bronchoscopic simulator (ORSIM) for 60 minutes before the subjects perform the 2nd Fiber optic intubation
  Arms: Simulator arm

SUMMARY:
The aim of the study is to study whether training by residents or anesthesia assistants, on a recently introduced virtual-reality bronchoscopic simulator (ORSIM) improves performance of fiberoptic intubation in patients.

DETAILED DESCRIPTION:
Traditionally, fiber optic bronchoscopy (FOB) intubation has been taught in a see one, do one basis. Modern training method in skill acquisition involves the use of simulators. Recently a portable, computer based, bronchoscopic simulator (ORSIM) was developed. The investigators hypothesized that operators trained with the ORSIM simulator will be more proficient in performing asleep FOB intubation than those trained with didactic teaching alone.

This randomized trial involves 34 consented residents or anesthesia assistants (AAs). In preparation, each consented person will view a teaching video of FOB intubation and tips. They will then perform an asleep FOBI in the OR under a staff anesthesiologist's supervision who's familiar with the study. Those who are randomized to the ORSIM group with undergo simulator training of 30-60 min. Those in the Didactic group will not undergo further training. Within about a week, the resident/AA will perform another asleep FOB intubation.

The study results will impact on how FOB intubation will be taught effectively in the future.

ELIGIBILITY:
Inclusion Criteria:

Subject:

* anesthesia/surgery/emergency/critical care residents or anesthesia assistants who have performed less than 5 Fiberoptic intubations

Exclusion Criteria:

* experience with bronchoscopy simulator or 5 or more FOB intubations

Patient:

* Anticipated difficult airway
* Mallampati Grade (MPG) >III
* Body Mass Index (BMI) >30

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Performance of Fiberoptic intubation assessed by validated 40 point Global Rating Scale (GRS) | 1 year

SECONDARY OUTCOMES:
Success/Failure of Fiberoptic intubation | 1 year
The duration (in seconds) of the Fiberoptic intubation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: David T Wong, MD, Principal Investigator — Department of Anesthesiology, Toronto Western Hospital, 399, Bathurst St., MC2-405, Toronto, ON, Canada M5T 1S8
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Wong DT, Mehta A, Singh KP, Leong SM, Ooi A, Niazi A, You-Ten E, Okrainec A, Patel R, Singh M, Wong J. The effect of virtual reality bronchoscopy simulator training on performance of bronchoscopic-guided intubation in patients: A randomised controlled trial. Eur J Anaesthesiol. 2019 Mar;36(3):227-233. doi: 10.1097/EJA.0000000000000890. PMID 30234669